CLINICAL TRIAL: NCT00169104
Title: A Phase II Trial of Trastuzumab, Neupogen, and Vinorelbine Investigating the Effects on Immune Function and Clinical Outcomes in Patients With Metastatic Breast Cancer Overexpressing Her-2/Neu
Brief Title: Effects of Granulocyte Colony-stimulating Factor (G-CSF), Trastuzumab, and Vinorelbine on Immune Cell Function
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Closed due to achievement of primary study endpoint
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Gary Schwartz, Staff Physician, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D-0140
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Results first posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-06

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast cancer; Her-2/neu; Granulocyte Colony Stimulating Factor; Trastuzumab; Vinorelbine; Antibody-dependent cellular cytotoxicity; Effector cells
MeSH Terms: conditions — Breast Neoplasms | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; Trastuzumab; Vinorelbine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Subjects will receive ten doses of G-CSF at a dose of 5 mcgm/kg daily Monday through Friday for the first two weeks of the trial. All patients will also receive trastuzumab at 4 mg/kg week 1, and 2 mg/kg week 2 during the first two weeks of the trial. All patients will then receive 12 weeks of trastuzumab at 2 mg/kg IV weeks 3 through 14, vinorelbine at 25 mg/m2 IV weekly weeks 3,4,6,7,9,10,12,13 and G-CSF at 5 mcgm/kg SQ daily Monday through Friday weeks 3-14.
  Interventions: Drug: G-CSF; Drug: trastuzumab; Drug: vinorelbine
- 2 (Placebo Comparator): Subjects will receive ten doses of a placebo injection SQ daily Monday through Friday for the first two weeks of the trial. All patients will also receive trastuzumab at 4 mg/kg week 1, and 2 mg/kg week 2 during the first two weeks of the trial. All patients will then receive 12 weeks of trastuzumab at 2 mg/kg weeks 3-14, vinorelbine at 25 mg/m2 IV weekly weeks 3,4,6,7,9,10,12,13, and G-CSF at 5 mcgm/kg SQ daily Monday through Fridays weeks 3-14.
  Interventions: Drug: G-CSF; Drug: trastuzumab; Drug: vinorelbine; Drug: saline placebo

INTERVENTIONS:
Drug: G-CSF — 5 mcgm/kg daily Monday through Friday weeks 3-14
  Other Names: Neupogen
Drug: trastuzumab — 4 mcgm/kg intravenously (IV) over 90 minutes week 1, then 2 mg/kg IV over 30 minutes weeks 2-14
  Other Names: Herceptin
Drug: vinorelbine — 25 mg/m2 over 6 minutes IV weekly, weeks 3, 4, 6, 7, 9, 10, 12, 13
  Other Names: Navelbine
Drug: G-CSF — 5 mcgm/kg SQ daily for ten days, Monday through Friday of the first two weeks of the study
  Other Names: Neupogen
  Arms: 1
Drug: saline placebo — Saline will be given SQ daily for ten days, Monday through Friday of the first two weeks of the study
  Arms: 2

SUMMARY:
Trastuzumab or Herceptin is an antibody directed against Her-2. Her-2 is a growth factor receptor which is present on the tumors of 25% of patients with breast cancer. The addition of trastuzumab to chemotherapy has been shown in a randomized clinical trial to increase the response rate to chemotherapy, the duration of response to chemotherapy, and to improve the duration of survival of patients with metastatic breast cancer. The anticancer mechanism of action of trastuzumab is unknown, but it is possible that trastuzumab acts by promoting antibody-dependent cell mediated cytotoxicity (ADCC), or direct killing of cancer cells by immune cells, triggered by antibodies bound to the surface of the cancer cell. G-CSF is a drug which is a growth factor for certain types of immune cells. G-CSF has two favorable effects on ADCC. G-CSF increases the pool of circulating cancer-killing immune cells, and G-CSF increases the strength of binding of cancer-killing immune cells to a specific part of the antibody. Therefore, priming with G-CSF significantly increases the efficiency of ADCC, and four days of treatment with G-CSF has been shown to optimize ADCC in some studies. Recent data from the investigators' laboratory indicates that chemotherapy can augment ADCC directed against tumor cells.

The investigators' hypothesis is that pre-treatment with the drug G-CSF would increase the effectiveness of chemotherapy given with trastuzumab.

DETAILED DESCRIPTION:
This is a randomized phase II study comparing trastuzumab with G-CSF against trastuzumab with placebo during the first two weeks of therapy.

Twenty five patients with metastatic breast cancer will be randomized to receive weekly trastuzumab plus either G-CSF or placebo by subcutaneous (SQ) injection daily for five days weekly for two weeks. Subsequently, all patients will receive an additional 12 weeks of weekly trastuzumab, G-CSF by SQ injection daily for five days weekly for 12 weeks, and vinorelbine once weekly at a dose of 25 mg/m2 weeks 3, 4, 6, 7, 9, 10, 12, 13. Baseline evaluation will include a history and physical exam, comprehensive metabolic panel (CMP), complete blood count (CBC), serum pregnancy test, computerized tomography (CT) scan for disease measurements, and a Multiple Uptake Gated Acquisition (MUGA) scan. The CT scan and MUGA will be repeated upon completion of the study treatment. Blood will be drawn pre-trastuzumab, 2 hours post-trastuzumab, and 48 hours post-trastuzumab on weeks 1, 2, 3, 4, and 12 to measure whole blood ADCC activity. Two additional assays for whole blood ADCC activity will be drawn at baseline pre-treatment, and following completion of protocol treatment. These assays will measure chromium release from a Her-2 positive target cell exposed to the patient's effector cells. Measurement of soluble Her-2 in patient serum will also be measured at each ADCC time point.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have pathological confirmation of carcinoma of the breast.
* Patients must have metastatic breast cancer by documented clinical or radiological assessment.
* Immunohistochemical analysis of HER-2/neu expression on paraffin-embedded specimens will be performed. HER-2/neu overexpression will be qualitatively scored as 0, 1+, 2+, or 3+, with 3+ indicating the strongest positivity. Fluorescence In Situ Hybridization (FISH) analyses will also be performed on these patients. Patients with 2+ to 3+ overexpression of HER-2/neu (membranous staining) are eligible, regardless of the results of the FISH analysis.
* Age ≥18 years.
* Karnofsky performance status ≥ 60%.
* Adequate hepatic, renal, and hematologic function.
* Prior treatment with trastuzumab will be allowed.
* All patients must have adequate cardiac function (defined as left ventricular ejection fraction ≥ 45%) documented by echocardiogram or MUGA scan.
* Premenopausal women will be required to have a negative urine or serum pregnancy test and to use an effective form of contraception.
* Patients with a history of brain metastases are permitted as long as it has been at least 30 days since definitive treatment, they are clinically stable and a magnetic resonance imaging scan of the brain demonstrates control of the lesion(s).
* All patients must give written informed consent indicating they are aware of the investigational nature of this treatment, as well as the risks and benefits of this protocol.

Exclusion Criteria:

* No treatment with chemotherapy or trastuzumab will be allowed within four weeks of study entry.
* Prior therapy with vinorelbine.
* Known history of hypersensitivity to trastuzumab, Chinese hamster ovary (CHO) cell proteins, or any component of these products.
* History of current unstable angina, symptomatic congestive heart failure, or myocardial infarction within the last 6 months.
* Pregnant women are excluded.
* History of a known hypersensitivity to E. coli-derived proteins, filgrastim, or any component of the product.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2002-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary N Schwartz, MD, Principal Investigator — Norris Cotton Cancer Center

REFERENCES:
- [Result] Schwartz GN, Kaufman PA, Tretter CPG, Arrick BA, Mulrooney TJ, Connelly EM, Mellinger DL, Fisher JL, Ernstoff MS. Vinorelbine and trastuzumab enhance effector cell function in patients with Her-2/neu overexpressing metastatic breast cancer. Breast Cancer Research and Treatment 88 (Suppl 1):S128a, 2004.
- See also: Norris Cotton Cancer Center Home Page — http://cancer.dartmouth.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between July 12, 2002 and November 2, 2007 from the Comprehensive Breast Program at the Norris Cotton Cancer Center.
Pre-assignment Details: There was no run-in prior to randomization and the start of treatment.
Groups:
- G-CSF Arm: Subjects will receive ten doses of G-CSF at a dose of 5 mcgm/kg daily Monday through Friday for the first two weeks of the trial. All patients will also receive trastuzumab at 4 mg/kg week 1, and 2 mg/kg week 2 during the first two weeks of the trial. All patients will then receive 12 weeks of trastuzumab at 2 mg/kg IV weeks 3 through 14, vinorelbine at 25 mg/m2 IV weekly weeks 3,4,6,7,9,10,12,13 and G-CSF at 5 mcgm/kg SQ daily Monday through Friday weeks 3-14.
- Placebo Arm: Subjects will receive ten doses of a placebo injection SQ daily Monday through Friday for the first two weeks of the trial. All patients will also receive trastuzumab at 4 mg/kg week 1, and 2 mg/kg week 2 during the first two weeks of the trial. All patients will then receive 12 weeks of trastuzumab at 2 mg/kg weeks 3-14, vinorelbine at 25 mg/m2 IV weekly weeks 3,4,6,7,9,10,12,13, and G-CSF at 5 mcgm/kg SQ daily Monday through Fridays weeks 3-14.
Period: Overall Study
Arm/Group | G-CSF Arm | Placebo Arm
Started | 13 | 10
Completed | 11 | 8
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: A total of 23 subjects were enrolled. Four subjects dropped out in the first week of treatment and are inevaluable for any study endpoints.
Groups:
- Total: Total of all reporting groups
Arm/Group | G-CSF Arm | Placebo Arm | Total
Number analyzed (Participants) | 11 | 8 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 7 | 17
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (10.0) | 53.9 (12.6) | 52.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Antibody Dependent Cell-mediated Cytotoxicity of Effector Cells Isolated From Subjects Receiving Trastuzumab With Either G-CSF or a Saline Placebo Against a Her-2 Overexpressing Target in Vitro
Description: Buffy coat effector cells were isolated by centrifugation from heparinized blood, and washed and counted. SKBR3 target cells were labeled with 51-Cr at 100 uCi per 5 x 105 cells for 1 hour at 37 C, washed and effector cells and target cells were plated at a ratio of 70:1 in 96 well microtiter plates, with trastuzumab 2 ug/ml and with no antibody. After addition of the target cells, the plate was centrifuged gently at 1200 rpm to pellet cells, the plate was incubated for 4 hours at 37C, and 100 uL of supernatant was measured on a gamma counter set for 51Cr counting for 1 minute per tube. Specific lysis in % is defined as follows:
  % specific lysis = (counts released into the supernatant under experimental conditions - spontaneous counts released into the supernatant) / (maximum counts released into the supernatant - spontaneous counts released into the supernatant)
  Specific lysis at Day 12 was compared to specific lysis at baseline between the G-CSF group and the placebo group.
Time Frame: Baseline and 12 days
Population: 19 subjects were evaluable for response and toxicity, but only 17 subjects had evaluable specific lysis laboratory outcomes at baseline and at Day 12.
Measure: Mean (Standard Deviation); unit: percentage of specific lysis
Groups:
- G-CSF Arm: Subjects will receive ten doses of G-CSF at a dose of 5 mcgm/kg daily Monday through Friday for the first two weeks of the trial. All patients will also receive trastuzumab at 4 mg/kg week 1, and 2 mg/kg week 2 during the first two weeks of the trial. All patients will then receive 12 weeks of trastuzumab at 2 mg/kg IV weeks 3 through 14, vinorelbine at 25 mg/m2 IV weekly weeks 3,4,6,7,9,10,12,13 and G-CSF at 5 mcgm/kg SQ daily Monday through Friday weeks 3-14.
  G-CSF: 5 mcgm/kg daily Monday through Friday weeks 3-14
  trastuzumab: 4 mcgm/kg intravenously (IV) over 90 minutes week 1, then 2 mg/kg IV over 30 minutes weeks 2-14
  vinorelbine: 25 mg/m2 over 6 minutes IV weekly, weeks 3, 4, 6, 7, 9, 10, 12, 13
  G-CSF: 5 mcgm/kg SQ daily for ten days, Monday through Friday of the first two weeks of the study
- Placebo Arm: Subjects will receive ten doses of a placebo injection SQ daily Monday through Friday for the first two weeks of the trial. All patients will also receive trastuzumab at 4 mg/kg week 1, and 2 mg/kg week 2 during the first two weeks of the trial. All patients will then receive 12 weeks of trastuzumab at 2 mg/kg weeks 3-14, vinorelbine at 25 mg/m2 IV weekly weeks 3,4,6,7,9,10,12,13, and G-CSF at 5 mcgm/kg SQ daily Monday through Fridays weeks 3-14.
  G-CSF: 5 mcgm/kg daily Monday through Friday weeks 3-14
  trastuzumab: 4 mcgm/kg intravenously (IV) over 90 minutes week 1, then 2 mg/kg IV over 30 minutes weeks 2-14
  vinorelbine: 25 mg/m2 over 6 minutes IV weekly, weeks 3, 4, 6, 7, 9, 10, 12, 13
  saline placebo: Saline will be given SQ daily for ten days, Monday through Friday of the first two weeks of the study
Arm/Group | G-CSF Arm | Placebo Arm
Number analyzed (Participants) | 10 | 7
percentage of specific lysis | 1.47 (0.97) | 1.67 (2.34)
Statistical Analysis 1: Comparison: G-CSF Arm vs Placebo Arm; T test; Test type: Superiority; p > 0.05, t-test, 2 sided — t=-0.29; df=15; Mean Difference (Net) = -0.20

2. Secondary Outcome: Antibody Dependent Cell-mediated Cytotoxicity of Effector Cells Isolated From Subjects Receiving Chemotherapy, Trastuzumab, and G-CSF Against a Her-2 Overexpressing Target in Vitro
Description: Buffy coat effector cells were isolated by centrifugation from heparinized blood, washed, and counted. SKBR3 target cells were labeled with 51-Cr at 100 uCi per 5 x 105 cells for 1 hour at 37 C, washed and effector cells and target cells were plated at a ratio of 70:1 in 96 well microtiter plates, with trastuzumab 2 ug/ml and with no antibody. After addition of the target cells, the plate was centrifuged gently at 1200 rpm to pellet cells, the plate was incubated for 4 hours at 37C, and 100 uL of supernatant was measured on a gamma counter set for 51Cr counting for 1 minute per tube. Specific lysis in % is defined as follows:
  % specific lysis = (counts released into the supernatant under experimental conditions - spontaneous counts released into the supernatant) / (maximum counts released into the supernatant - spontaneous counts released into the supernatant)
  Specific lysis at Week 14 was compared to specific lysis at baseline for 17 patients with week 14 samples available.
Time Frame: Baseline and 14 weeks
Population: 17 of 19 subjects had results from ADCC assays from baseline and at week 14. Because subjects on both arms of the trial received the identical treatment with 12 weeks of vinorelbine and G-CSF after the initial two week randomization, it is appropriate to pool the results of the ADCC assays at the 14 week timepoint from both arms.
Measure: Median (Standard Deviation); unit: percentage of specific lysis
Arm/Group | All Patients
Number analyzed (Participants) | 17
percentage of specific lysis | 1.67 (3.47)

3. Secondary Outcome: Clinical Response Rate of the Combination of Trastuzumab, G-CSF, and Vinorelbine in Subjects With Her-2 Overexpressing Metastatic Breast Cancer
Description: 19 subjects (11 on the G-CSF arm and 8 on the placebo arm) completed 14 weeks of treatment and completed restaging at that time.
  Responses were evaluated by RECIST criteria.
Time Frame: 14 weeks
Population: 19 subjects completed 14 weeks of treatment and underwent restaging at that timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | G-CSF Arm | Placebo Arm
Number analyzed (Participants) | 11 | 8
Participants
  Complete Response | 0 | 0
  Partial Response | 1 | 4
  Stable Disease | 2 | 3
  Disease Progression | 8 | 1

4. Secondary Outcome: Safety of the Combination of Trastuzumab, G-CSF, and Vinorelbine in Subjects With Her-2 Overexpressing Metastatic Breast Cancer
Description: Adverse events were graded per RECIST v4.0. There were two severe adverse events: Grade 3 mental status changes in one subject on the G-CSF arm, and Grade 3 febrile neutropenia in one subject on the Placebo arm.
  Refer to Adverse Events Table for specifics.
Time Frame: 14 weeks
Population: 19 subjects (11 on the G-CSF arm and 8 on the placebo arm) received at least two weeks of treatment on study and were evaluable for toxicity.
Measure: Count of Participants; unit: Participants
Arm/Group | G-CSF Arm | Placebo Arm
Number analyzed (Participants) | 11 | 8
Participants
  Grade 3 mental status changes | 1 | 0
  Grade 3 febrile neutropenia | 0 | 1
  Grade 4 leukopenia | 2 | 0
  Grade 4 granulocytopenia | 1 | 0
  Grade 3 anemia | 3 | 0
  Grade 3 thrombocytopenia | 1 | 0
  Grade 3 granulocytopenia | 2 | 1
  Grade 3 elevation in alkaline phosphatase | 2 | 1
  Grade 3 elevation in AST | 1 | 0
  Grade 3 elevation in ALT | 0 | 1
  Grade 2 sensory neuropathy | 1 | 1
  Grade 2 arthralgias | 0 | 2
  Grade 2 constipation | 1 | 1
  Grade 2 tumor pain | 0 | 1
  Grade 2 mucositis | 0 | 1
  Grade 2 heartburn | 1 | 0
  Grade 2 anemia | 5 | 4
  Grade 2 thrombocytopenia | 0 | 1
  Grade 2 leukopenia | 3 | 1
  Grade 2 granulocytopenia | 1 | 1
  Grade 2 elevation in alkaline phosphatase | 5 | 2
  Grade 2 elevation in AST | 0 | 2
  Grade 2 elevation in ALT | 0 | 1

ADVERSE EVENTS:
Time Frame: 14 weeks
Groups:
- G-CSF: Subjects will receive ten doses of G-CSF at a dose of 5 mcgm/kg daily Monday through Friday for the first two weeks of the trial. All patients will also receive trastuzumab at 4 mg/kg week 1, and 2 mg/kg week 2 during the first two weeks of the trial. All patients will then receive 12 weeks of trastuzumab at 2 mg/kg IV weeks 3 through 14, vinorelbine at 25 mg/m2 IV weekly weeks 3,4,6,7,9,10,12,13 and G-CSF at 5 mcgm/kg SQ daily Monday through Friday weeks 3-14.
  G-CSF: 5 mcgm/kg daily Monday through Friday weeks 3-14
  trastuzumab: 4 mcgm/kg intravenously (IV) over 90 minutes week 1, then 2 mg/kg IV over 30 minutes weeks 2-14
  vinorelbine: 25 mg/m2 over 6 minutes IV weekly, weeks 3, 4, 6, 7, 9, 10, 12, 13
  G-CSF: 5 mcgm/kg SQ daily for ten days, Monday through Friday of the first two weeks of the study
- {Placebo: Subjects will receive ten doses of a placebo injection SQ daily Monday through Friday for the first two weeks of the trial. All patients will also receive trastuzumab at 4 mg/kg week 1, and 2 mg/kg week 2 during the first two weeks of the trial. All patients will then receive 12 weeks of trastuzumab at 2 mg/kg weeks 3-14, vinorelbine at 25 mg/m2 IV weekly weeks 3,4,6,7,9,10,12,13, and G-CSF at 5 mcgm/kg SQ daily Monday through Fridays weeks 3-14.
  G-CSF: 5 mcgm/kg daily Monday through Friday weeks 3-14
  trastuzumab: 4 mcgm/kg intravenously (IV) over 90 minutes week 1, then 2 mg/kg IV over 30 minutes weeks 2-14
  vinorelbine: 25 mg/m2 over 6 minutes IV weekly, weeks 3, 4, 6, 7, 9, 10, 12, 13
  saline placebo: Saline will be given SQ daily for ten days, Monday through Friday of the first two weeks of the study
Arm/Group | G-CSF | {Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/11 | 1/8
Other Adverse Events (participants affected / at risk) | 10/11 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-CSF (N=11) | {Placebo (N=8)
Mental status change (Nervous system disorders) | 1 (1) | 0 (0) — Grade 3
Febrile neutropenia (Immune system disorders) | 0 (0) | 1 (1) — Grade 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | G-CSF (N=11) | {Placebo (N=8)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Grade 3
Anemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) — Grade 3
Sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1) — Grade 2
Arthralgias (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) — Grade 2
constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) — Grade 2
anemia (Blood and lymphatic system disorders) | 5 (5) | 4 (4) — Grade 2
Tumor pain (Nervous system disorders) | 0 (0) | 1 (1) — Grade 2
Mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 2
heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Grade 2
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Grade 4
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) — Grade 2
Granulocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Grade 4
Granulocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) — Grade 3
Granulocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — Grade 2
Elevated alkaline phosphatase (Investigations) | 2 (2) | 1 (1) — Grade 3
Elevated alkaline phosphatase (Investigations) | 5 (5) | 2 (2) — Grade 2
Elevated AST (Investigations) | 1 (1) | 0 (0) — Grade 3
Elevated AST (Investigations) | 0 (0) | 2 (2) — Grade 2
Elevated ALT (Investigations) | 0 (0) | 1 (1) — Grade 3
Elevated ALT (Investigations) | 0 (0) | 1 (1) — Grade 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor will be provided 30 days to review a manuscript and 15 days to review a poster. The sponsor may request an additional 60 days to review study results prior to their release, if the request is submitted in writing.